CLINICAL TRIAL: NCT05312112
Title: Real World Outcomes Using Novel Agents for Acute Myeloid Leukaemia in the United Kingdom
Brief Title: Real World Outcomes Using Novel Agents for AML in the UK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 305432; 305432 (Other: IRAS)
Record Dates: First submitted 2022-03-09; First posted 2022-04-05 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; gilteritinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Venetoclax: Venetoclax in newly diagnosed AML
  Interventions: Drug: Venetoclax
- FLT3 inhibitors: FLT3 inhibitors including gilteritinib in relapsed AML
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Venetoclax — Observational study of venetoclax in AML
  Other Names: Venclyxto
  Groups: Venetoclax
Drug: Gilteritinib — Observational study of gilteritinib in AML
  Other Names: Xospata
  Groups: FLT3 inhibitors

SUMMARY:
This project will collect data on patients with acute myeloid leukemia in the United Kingdom who were treated with two new targeted therapies during the coronavirus pandemic

DETAILED DESCRIPTION:
Acute myeloid leukaemia (AML) is a blood cancer which in fit young adults is typically treated with intensive chemotherapy. While this is potentially curative, it is associated with significant side effects and the requirement for long hospital admissions. Infection is a major issue during AML treatment, as both the disease and the chemotherapy impair the immune system.

Early data suggested that COVID-19 is associated with a very high rate of death in AML patients undergoing intensive chemotherapy. Because of this, and the need for significant hospital resources to deliver intensive chemotherapy, the NHS made available two new, less intensive, targeted therapies for the treatment of AML during the COVID-19 pandemic - venetoclax and gilteritinib. The aim was to reduce mortality and healthcare resource use.

Many hundreds of patients across the UK have been treated with these two medications on the temporary access scheme. The research aims to collect de-identified data from treating patients to describe the outcomes of patients treated with these approaches, both in terms of the safety and effectiveness.

ELIGIBILITY:
Venetoclax cohort Inclusion criteria

1. Newly diagnosed acute myeloid leukaemia
2. No prior therapies for AML, apart from hydroxyurea (or similar) for cytoreduction. Previous treatments for MDS or other conditions are allowed
3. Treated with venetoclax in combination with either azacitidine or LDAC No exclusion criteria

Gilteritinib/FLT3 cohort Inclusion criteria

1. Relapsed acute myeloid leukaemia, including molecular relapse
2. Treated with FLT3 inhibitor No exclusion criteria

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The NHS criteria for access to venetoclax was that a patient was fit for IC and was:
  * Aged >16y with NPM1 mutation without FLT3 internal tandem duplication (ITD)
  * Aged >50y with NPM1, IDH1 or IDH2 mutations (regardless of FLT3 status)
  * Patients aged >60y without favourable-risk cytogenetics
  Gilteritinib was made available to all patients aged >16y with relapse or refractory FLT3 mutated AML. Other FLT3 inhibitors are available to patients through various access schemes
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Overall survival measured from time of treatment initiation
Early death rate | Day 60 after starting treatment
  Early death rate measured at day 60 after treatment initiation

SECONDARY OUTCOMES:
Response rate | After 2 cycles of therapy (each cycle is 28 days although may be extended if recovery is delayed)
  Response rate as defined by ELN 2017
Incidence of relapse in patients achieving remission | 1 year
  Relapse incidence measured from the time of achieving remission
Relapse-free survival | 1 year
  RFS as defined by ELN
Treatment toxicity 1 | During the first cycle of therapy (each cycle is 28 days although may be extended if recovery is delayed)
  Number of days in hospital and number of days of intensive care
Treatment toxicity 2 | During the first cycle of therapy (each cycle is 28 days although may be extended if recovery is delayed)
  Duration of neutropenia and thrombocytopenia
Treatment toxicity 3 | During the first cycle of therapy (each cycle is 28 days although may be extended if recovery is delayed)
  Number of blood and platelet transfusions
Comparison of survival between patient sub-groups | 1 year
  Overall survival compared between disease groups

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dillon, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided